CLINICAL TRIAL: NCT07312110
Title: D-SPARK: A Randomized Double Blind Clinical Trial of D-Serine for Modifying Parkinson's Disease Progression
Brief Title: D-SPARK: A Clinical Trial of D-Serine for Modifying Parkinson's Disease Progression
Acronym: D-SPARK
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Haukeland University Hospital (Other)
Collaborators: SPARK NS (Unknown); University of Bergen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: REK: 929216
Record Dates: First submitted 2025-11-21; First posted 2025-12-31 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2026-01

CONDITIONS: Parkinson s Disease; Parkinson Disease (PD)
Keywords: Serine; Parkinsons disease; D-serine
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Intervention Model Description: All participants will be assigned to placebo and D-serine at different time periods during the course of the study.
Who Masked: Participant, Care Provider, Investigator
Masking Description: Double-blinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Early-start (Active Comparator): Participants in this group will receive D-serine at an earlier time point than the placebo group. All participants will receive placebo and D-serine at different parts of the study.
  Interventions: Dietary Supplement: D-serine; Dietary Supplement: Placebo
- Delayed-start (Placebo Comparator): Participants in this group will receive D-serine at a later time point than the early-start group. All participants will receive placebo and D-serine at different parts of the study
  Interventions: Dietary Supplement: D-serine; Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: D-serine — D-serine 2 x 500 mg and 2 x Placebo oral capsules administered twice daily the first week of intervention, then uptitrated to D-serine 4 x 500 mg twice daily for the remainder of the intervention.
Dietary Supplement: Placebo — Placebo 2 x oral capsules administered twice daily.

SUMMARY:
This clinical study, designed as a randomized, double-blind, placebo-controlled trial, aims to investigate if modulation of the N-methyl-D-aspartate receptor (NMDAR) via its co-agonist D-serine has therapeutic benefits in Parkinson's disease (PD). All patients will receive both placebo and D-serine over different time periods during the study.

Preclinical studies have shown that blocking glycine transporters, which elevates endogenous glycine levels, can restore NMDAR function and improve motor deficits in PD models. A clinical trial demonstrated that oral D-serine (30 mg/kg/day for 6 weeks) significantly reduced extrapyramidal and abnormal involuntary movements in PD patients compared to placebo, with improvements observed in both motor and non-motor symptoms. D-serine supplementation has shown an acceptable safety profile with doses up to 120 mg/kg showing no significant adverse effects in clinical studies.

The D-SPARK trial primarily aims to determine the efficacy of D-serine supplementation on clinical severity of PD as measured by the Movement Disorder Society Unified Parkinson's Disease Rating Scale (MDS-UPDRS).

Secondary aims are to determine the efficacy of D-serine supplementation on improving dopaminergic nigrostriatal innervation as measured by single-photon emission tomography (SPECT) based imaging of the dopamine transporter (DaT-scan) and cognition as measured by the California Verbal Learning Test version 2 (CLVT-II).

The study will include 100 persons with Parkinson's disease (PwPD) diagnosed no longer than 5 years before baseline. Participants will be randomly assigned to receive D-Serine 4000 mg daily or placebo for defined periods of time during a 58 week treatment period, followed by a 12 week washout period.

Participants will undergo:

* Clinical evaluations, including clinical rating scales and questionnaires.
* Cognitive assessments.
* Bio sampling of whole blood and blood plasma.
* Single-photon emission tomography (SPECT) imaging of dopamine transporter levels (DaT-scan)

The outcomes of this study could potentially demonstrate that D-serine reduces symptom severity in Parkinson's disease and/or has an impact on the clinical trajectory of Parkinson's disease, benefiting persons living with Parkinson's disease, their families and society as a whole.

DETAILED DESCRIPTION:
The study design is a randomized, double-blind, placebo-controlled trial.

The trial consists of 3 stages followed by a washout period.

* Screening and antiparkinsonian treatment optimization:

  --- Potential participants will be screened for eligibility and consented for participation. Treatment of Parkinson's disease with dopaminergic drugs will be initiated/adjusted until an optimal, stable effect of treatment is established. This treatment regimen will be maintained throughout the first 32 weeks of the intervention stage, after which changes will be allowed. If an optimal, stable dose is not achieved during screening, these participants will not proceed further and will not be included in the study.
* Intervention stage:

  --- Participants will undergo randomization and will be assigned to receive either placebo or D-serine during different portions of the intervention phase. Participants will receive study drug (placebo or D-serine) for a total of 58 weeks. Thirty-two weeks after starting study drug, participants may have their dopaminergic drugs adjusted, if necessary.
* Washout stage:

  * Upon completion of the intervention period, participants will discontinue study drug and will be followed for an additional 12 weeks. A final study visit will occur 12 weeks after discontinuation of study drug.

ELIGIBILITY:
Inclusion Criteria:

* A clinical diagnosis of PD* according to the clinically established MDS clinical diagnostic criteria for Parkinson's disease within 5 years.
* [¹²³I]FP-CIT single photon emission CT (DaTscan) confirming dopaminergic nigrostriatal denervation.
* Hoehn and Yahr score < 3 at enrollment.
* Optimal symptomatic PD treatment, not requiring adjustments, for at least 2 weeks.
* Age ≥40 and ≤ 80 years at time of enrollment.

Exclusion Criteria:

* Dementia or neurodegenerative disorder other than PD at baseline visit.
* Atypical parkinsonism (PSP, MSA, CBD vascular parkinsonism, or drug induced parkinsonism).
* Any known monogenic cause of PD (GBA1 variation is accepted).
* Any psychiatric disorder that would interfere with compliance in the study.
* Any severe somatic illness that would make the individual unable to comply and participate in the study.
* Use of D-serine supplementation within 90 days of enrolment.
* Metabolic, neoplastic, or other physically or mentally debilitating disorder at baseline visit.
* Active of planned pregnancy during trial period.
* Cognitive impairment as measured by the Mini Mental Status Exam MMSE) < 20.
* Weight < 45 kg.
* Urinary albumin/creatinine ratio ≥ 20 mg/mmol at time of enrollment.
* Participants will be excluded if they have CKD stage 3 or higher, defined as:

  * Estimated golumerular filtration rate (eGFR) < 60 mL/min/1.73min^2 at screening, calculated using the CKD-EPI 2021 creatinine equation.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2028-03 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Change in MDS-UPDRS Total Score (sum of Parts I-III). | 26 weeks.
  Difference between treatment groups (DSR vs placebo) in mean change from baseline to Week 26 in Movement Disorder Society Unified Parkinson's Disease Rating Scale (MDS-UPDRS) Total Score (sum of Parts I-III), assessed in all randomized participants under a treatment-policy strategy. MDS-UPDRS Part III tested in the OFF-medication state.
  MDS-UPDRS sum of part I-III: Clinical rating scale of motor and non-motor symptoms of Parkinson's Disease. Part I (13 items; Score 0-52) examines non-motor experiences, Part II (13 items; Score 0-52) examines motor experiences of daily living, Part III (33 items; Score 0-132) examines the cardinal motor disabilities. Each Part has 0-4 ratings, where 0 (no problems) to 4 (severe problems) and scores for each part are summed to calculate the total score which ranges from 0-236. Higher scores represent a worse outcome.

SECONDARY OUTCOMES:
Change in mean striatal binding ratio (SBR) of the putamen bilaterally, measured by [¹²³I] FP-CIT Single-Photon Emission Computed Tomography (SPECT) Imaging of the Dopamine Transporter (DaT-scan). | 26 Weeks.
  Difference between treatment groups (DSR vs Placebo) in mean change from baseline to Week 26 in the mean striatal binding ratio (SBR) of the putamen, bilaterally, as measured by [¹²³I] FP-CIT Single-Photon Emission Computed Tomography (SPECT) Imaging of the Dopamine Transporter (DaT-scan). Assessed in all randomized participants under a treatment-policy strategy.
Change in MDS-UPDRS part III score. | 26 Weeks.
  Difference between treatment groups (DSR vs placebo) in mean change from baseline to Week 26 in Movement Disorder Society Unified Parkinson's Disease Rating Scale (MDS-UPDRS) part III, assessed in all randomized participants under a treatment-policy strategy. MDS-UPDRS Part III tested in the OFF-medication state.
  MDS-UPDRS part III: Clinical rating scale of motor symptoms of Parkinson's Disease (33 items; Score 0-132). Higher scores represent worse outcomes.
Change in EQ-5D-5L index value. | 26 Weeks.
  Difference between treatment groups (DSR vs placebo) in mean change from baseline to Week 26 in the EQ-5D-5L index value, assessed in all randomized participants under a treatment-policy strategy. The scale measures quality of life on a 5-component scale with severity ranging from 0-5. An index from these is calculated based on country specific reference data and ranges from 0 to 1. Higher index score indicates a better outcome.
Change in CVLT-II total Score and sub-scores. | 26 Weeks.
  Difference between treatment groups (DSR vs placebo) in mean change from baseline to Week 26 in the California Verbal Learning Test version II (CVLT-II; Total Score and Sub-scores individually), assessed in all randomized participants under a treatment-policy strategy.
  CVLT-II: Verbal learning test assessing short delay and long delay recall and recognition. Separated into: Total score: Immediate Recall (sum of List A tests 1-5). Sub-scores: Short Delay Free Recall, Short Delay Cued Recall, Long Delay Free Recall, Long Delay Cued Recall, Long Delay Recognition, Forced Recognition.
  Higher CVLT-II scores indicate a better outcome.

OTHER OUTCOMES:
Change in MDS-UPDRS part I score. | 26 Weeks.
  Difference between treatment groups (DSR vs placebo) in mean change from baseline to Week 26 in Movement Disorder Society Unified Parkinson's Disease Rating Scale (MDS-UPDRS) part I, assessed in all randomized participants under a treatment-policy strategy. MDS-UPDRS is a Clinical rating scale of motor and non-motor symptoms of Parkinson's Disease. Part I (13 items; Score 0-52) examines non-motor experiences. Higher scores represent a worse outcome.
Change in MDS-UPDRS part II score. | 26 Weeks.
  Difference between treatment groups (DSR vs placebo) in mean change from baseline to Week 26 in Movement Disorder Society Unified Parkinson's Disease Rating Scale (MDS-UPDRS) part II, assessed in all randomized participants under a treatment-policy strategy.
  MDS-UPDRS part II: Clinical rating scale of motor experiences of daily living (13 items; Score 0-52). Higher scores indicate worse outcomes.
Change in MDS-UPDRS part IV score. | 26 Weeks.
  Difference between treatment groups (DSR vs placebo) in mean change from baseline to Week 26 in Movement Disorder Society Unified Parkinson's Disease Rating Scale (MDS-UPDRS) part IV, assessed in all randomized participants under a treatment-policy strategy.
  MDS-UPDRS part IV evaluates motor complications related to PD and contains 6 items scored by the clinician based on patient history from the preceding week (Range 0-24). Higher scores indicate a worse outcome.
Change in MoCA total score. | 26 Weeks.
  Difference between treatment groups (DSR vs placebo) in mean change from baseline to Week 26 in Montreal Cognitive Assessment (MoCA) Total Score, assessed in all randomized participants under a treatment-policy strategy.
  MoCA is a validated global measure of cognitive ability. Total score ranges from 0-30 with higher scores indicating a better outcome.
Change in Hoehn and Yahr Stage. | 26 Weeks.
  Difference between treatment groups (DSR vs placebo) in mean change from baseline to Week 26 in Hoehn and Yahr Stage, assessed in all randomized participants under a treatment-policy strategy.
  Hoehn and Yahr s cale distinguishes between five stages in PD, from unilateral impairment (Stage 1) to bilateral impairment without postural control difficulties, to postural instability (Stage 3), to severe disabling disease; still able to walk or stand unassisted (Stage 4) and finally Confinement to bed or wheelchair unless aided (Stage 5)
Change in B-SIT total score. | 26 weeks and 52 weeks.
  Difference between treatment groups (DSR vs placebo) in mean change from baseline to Week 26 and to Week 52 in the Brief Smell Identification Test (B-SIT) Total Score, assessed in all randomized participants under a treatment-policy strategy. The scale measures olfaction and has a range of 0-12, with higher scores indicating a better outcome.
Change in average walking-speed, measured using the Axivity Ax06 sensor. | 26 weeks and 52 weeks.
  Difference between treatment groups (DSR vs placebo) in mean change from baseline to Week 26 and to Week 52 in average walking-speed in m/s, assessed in all randomized participants under a treatment-policy strategy. Measured using the Axivity Ax06 accelerometer sensors placed on the wrist, lumbar back and thigh. Average walking-speed will be calculated as the mean walking-speed over a 7-day observation period before each study visit.
Change in blood/plasma levels of dopamine and related metabolite levels. | 26 weeks.
  Difference between treatment groups (DSR vs placebo) in mean change from baseline to Week 26 in blood/plasma dopamine and related metabolite levels, assessed in all randomized participants under a treatment-policy strategy.
Change in MDS-UPDRS parts I, II and III (Total and Sub-scores). | 52 weeks.
  Mean change from baseline within and between treatment groups (early-start and delayed-start) to Week 52 in Movement Disorder Society Unified Parkinson's Disease Rating Scale (MDS-UPDRS) Parts I, II, and III (Total and Sub-scores), assessed in all randomized participants under a treatment-policy strategy. MDS-UPDRS Part III tested in the OFF-medication state.
  MDS-UPDRS part I-III: Clinical rating scale of motor and non-motor symptoms of Parkinson's Disease. Part I (13 items; Score 0-52) examines non-motor experiences, Part II (13 items; Score 0-52) examines motor experiences of daily living, Part III (33 items; Score 0-132) examines the cardinal motor disabilities. Each Part has 0-4 ratings, where 0 (no problems) to 4 (severe problems) and scores for each part are summed to calculate the total score which ranges from 0-236. Higher scores represent a worse outcome.
Change in MDS-UPDRS Total Score (sum of parts I-III). | 52 weeks.
  Difference between treatment groups (early-start vs delayed start treatment groups) in mean change from baseline to Week 52 in Movement Disorder Society Unified Parkinson's Disease Rating Scale (MDS-UPDRS) Total Score (sum of parts I, II and III), assessed in all randomized participants under a treatment-policy strategy. MDS-UPDRS Part III tested in the OFF-medication state.
  MDS-UPDRS sum of parts I-III: Clinical rating scale of motor and non-motor symptoms of Parkinson's Disease. Part I (13 items; Score 0-52) examines non-motor experiences, Part II (13 items; Score 0-52) examines motor experiences of daily living, Part III (33 items; Score 0-132) examines the cardinal motor disabilities. Each Part has 0-4 ratings, where 0 (no problems) to 4 (severe problems) and scores for each part are summed to calculate the total score which ranges from 0-236. Higher scores represent worse outcomes for each part and total score.
Change in Levodopa Equivalent Daily Dose. | 26 weeks and 52 weeks.
  Difference between treatment groups (DSR vs Placebo) in mean change from baseline to Week 26 and Week 52 in Levodopa Equivalent Daily Dose (LEDD), assessed in all randomized participants under a treatment-policy strategy.
Change in serum inflammatory cytokine levels. | 26 weeks and 52 weeks.
  Difference between treatment groups (DSR vs placebo) in mean change from baseline to Week 26 and to Week 52 in serum cytokines, assessed in all randomized participants under a treatment-policy strategy. Serum cytokines include: TNF-a, IL-1b, IL-2, IL-6, IL-10, IFN-γ.
Change in neurofilament light chain levels. | 26 weeks and 52 weeks.
  Difference between treatment groups (DSR vs placebo) in mean change from baseline to Week 26 and to Week 52 in serum neurofilament light chain (NfL) levels, assessed in all randomized participants under a treatment-policy strategy.
Change in serum DSR levels. | 26 weeks and 52 weeks.
  Serum D-serine (DSR) levels at Week 26 and Week 52.
Change in MDS-UPDRS Toal Score (sum of parts I-III). | 64 weeks.
  Mean change from baseline within and between treatment groups (early-start and delayed-start) to Week 64 (12 weeks after IP discontinuation) in Movement Disorder Society Unified Parkinson's Disease Rating Scale (MDS-UPDRS) Total Score (sum of parts I, II and III), assessed in all randomized participants under a treatment-policy strategy. MDS-UPDRS Part III tested in the OFF-medication state.
  MDS-UPDRS sum of parts I-III: Clinical rating scale of motor and non-motor symptoms of Parkinson's Disease. Part I (13 items; Score 0-52) examines non-motor experiences, Part II (13 items; Score 0-52) examines motor experiences of daily living, Part III (33 items; Score 0-132) examines the cardinal motor disabilities. Each Part has 0-4 ratings, where 0 (no problems) to 4 (severe problems) and scores for each part are summed to calculate the total score which ranges from 0-236. Higher scores represent worse outcomes for each part and total score.
Change in CVLT-II Total Score and Sub-scores. | 64 weeks.
  Mean change from baseline within and between treatment groups (early-start and delayed-start) to Week 64 (12 weeks after IP discontinuation) in the California Verbal Learning Test version II (CLVT-II; Total Score and Sub-scores) and mean Montreal Cognitive Assessment (MoCA) Total Score, assessed in all randomized participants under a treatment-policy strategy.
  CVLT-II: Verbal learning test assessing short delay and long delay recall and recognition. Separated into: Total score: Immediate Recall (sum of List A tests 1-5). Sub-scores: Short Delay Free Recall, Short Delay Cued Recall, Long Delay Free Recall, Long Delay Cued Recall, Long Delay Recognition, Forced Recognition. Higher CVLT-II scores indicate a better outcome.
  MoCA is a validated global measure of cognitive ability. Total score ranges from 0-30 with higher scores indicating a better outcome.
Change in EQ-5D-5L index value. | 64 weeks.
  Mean change from baseline within and between treatment groups (early-start and delayed-start) to Week 64 (12 weeks after IP discontinuation) in the EQ-5D-5L index value, assessed in all randomized participants under a treatment-policy strategy. The scale measures quality of life on a 5-component scale with severity ranging from 0-5. An index from these is calculated based on country specific reference data and ranges from 0 to 1. Higher index score indicates a better outcome.
Frequency and severity of mild, moderate and severe adverse events (AE) and serious adverse events (SAE). | 64 weeks.
  Frequency and severity of mild, moderate, and severe Adverse Events and Serious Adverse Events occurring from 1st screening visit after participant has consented to study participation up to the end of study visit at Week 64 (12 weeks after discontinuation of IP). Classified as treatment-emerging if occurring after randomization.

CONTACTS AND LOCATIONS:
Locations (11):
- Norway (11):
  - Sørlandet Hospital Arendal, Arendal, Agder
  - Akershus University Hospital, Lørenskog, Akershus
  - Vestre Viken Hospital, Drammen, Buskerud
  - Molde Hospital, Molde, Møre og Romsdal
  - Bodø Hospital (Nordland Hospital), Bodø, Nordland
  - Oslo University Hospital, Oslo, Oslo County
  - Haugesund Hospital, Haugesund, Rogaland
  - University Hospital of North Norway, Tromsø, Troms
  - Haukeland University Hospital, Bergen, Vestland
  - Førde Hospital, Førde, Vestland
  - Østfold Hospital, Sarpsborg, Østfold fylke

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data in pseudonomized format will be shared with collaborators for analysis based on data tranfer agreements adhering to the Eu's General Data Protection Regulation (GDPR).